CLINICAL TRIAL: NCT04168788
Title: Pharmacogenetic Study of Antimitotic Therapies Involved in Hepatic Veno-occlusive Disease in Children With Nephroblastoma or Acute Lymphoblastic Leukemia
Brief Title: Pharmacogenetic Study of Antimitotic Therapies Involved in Hepatic VOD in Children With Nephroblastoma or ALL
Acronym: MVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 49RC19_0197
Record Dates: First submitted 2019-11-05; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Hepatic Veno-Occlusive Disease; Nephroblastoma; Acute Lymphoblastic Leukemia
Keywords: Pharmacogenetics
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease; Wilms Tumor; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Hematologic Tests; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nephrobalstoma or ALL (Other): Pateints treated for a nephrobalstoma or ALL in childhood or adolescence
  Interventions: Other: Blood test for genetic analysis

INTERVENTIONS:
Other: Blood test for genetic analysis — Drawing blood to realize a genetic analysis for susceptibility to hepatic VOD.

SUMMARY:
Hepatic veno-occlusive diseases (VOD) during cancer treatment in children are serious toxicities that have occurred with interruptions of chemotherapy and risk of relapse. In addition, these toxicities have a negative impact on the patient's quality of life, serious long-term sequelae and are potentially fatal in children.

The risk factors associated with the occurrence of these complications are, to date, unknown, at the exception to the exposition to certain treatments (6-thioguanine, busulfan, actinomycin D, radiotherapy, etc.). To understand the effects of this toxicity and those of susceptibility to the disease becomes a major issue in the treatment of these children.

DETAILED DESCRIPTION:
Case-control study, nested in two French multicenter cohorts, on pharmacognenetic, biological and clinical susceptibility factors associated with the occurrence of hepatic veno-occlusive disease during the anticancer treatment for nephroblastoma or acute lymphoblastic leukemia, with centralized genetic analysis.

After obtaining consent (patient or parents for minor patients), a blood sample is collected during the routine follow-up consultation and tubes are sent directly to Paris for the pharmacogenetic analysis at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged < 18 years old at the time of cancer diagnosis
* Having been treated with a single line of treatment for nephroblastoma or ALL, in France between 2000 and 2018, and who did not receive allogeneic hematopoietic stem cell transplantation
* Weight greater than 5 kg at inclusion
* Informed consent dated and signed by the holder of the parental authority (if minor) or by the patient (if major) to take part in the study
* Affiliated to a Social Security scheme

Exclusion Criteria:

* Unavaibility of constitutional DNA
* Person who receive more than one treatment line for nephroblastoma or ALL in childhood or adolescence
* Pregnant, lactating or parturient women
* Person deprived of their liberty by judicial or administrative decision
* Person under psychiatric care under duress
* Person subject to legal protection
* Person unable to express their consent

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlate pharmacogenetic analysis with veno-occlusive disease. | One day
  Illumina's "Human Omni2.5-8 v1.3" microarrays explore more than 2,600,000 genetic variants, thus covering the entire genome with more than 300,000 genetic biomarkers in exons.

SECONDARY OUTCOMES:
Participant characteristics. | One day
  Age, sociodemographics, personal and cancer history.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pellier, MD, Principal Investigator — University Hospital, Angers
Locations (16):
- France (16):
  - Univesity Hostipal of Amiens, Amiens
  - University Hospital of Bordeaux, Bordeaux
  - University of Brest, Brest
  - University Hospital of Dijon, Dijon
  - Centre Oscar Lambret, Lille
  - University Hospital of Limoges, Limoges
  - Hôpital La Timone, Marseille
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - Institut Curie, Paris
  - Hôpital Trousseau, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - University Hospital of La Réunion, Saint-Denis
  - University Hospital of Tours, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No